CLINICAL TRIAL: NCT04094376
Title: Comparison of Morning Operation and Evening Operation on Postoperative Sleep Quality and Pain Under General Anesthesia： A Randomized Controlled Trial
Brief Title: Comparison of Morning Operation and Evening Operation on Postoperative Sleep Quality and Pain Under General Anesthesia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shengjing Hospital (Other)
Responsible Party: Principal Investigator, Yanchao Yang, Principal investigator, Shengjing Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: circadian rhythm and sleep
Record Dates: First submitted 2019-09-17; First posted 2019-09-18 (Actual); Last update posted 2020-04-24 (Actual); Status verified 2020-04

CONDITIONS: Morning Operation; Evening Operation; Sleep Quality; General Anesthesia; Circadian Rhythm Sleep Disorder
Keywords: morning operation; evening operation; sleep quality; general anesthesia; circadian rhythm
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders; Sleep Disorders, Circadian Rhythm

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Day group (Other): 42 patients scheduled for elective laparoscopic abdominal surgeries under general anesthesia were randomly assigned to receive operation in the Day Group (8:00-12:00)
  Interventions: Other: receiving operation during the day or at night
- Night group (Other): 42 patients scheduled for elective laparoscopic abdominal surgeries under general anesthesia were randomly assigned to receive operation in the Night Group (18:00-22:00)
  Interventions: Other: receiving operation during the day or at night

INTERVENTIONS:
Other: receiving operation during the day or at night — eighty-four patients scheduled for elective laparoscopic abdominal surgeries under general anesthesia were randomly assigned to receive operation in the Day Group (8:00-12:00) and the Night Group (18:00-22:00)

SUMMARY:
General anesthesia is a medically induced state of low reactivity consciousness involving amnesia, immobility, unconsciousness, and analgesia, which is similar to natural sleep. Its aim is to create a state of sensory deprivation to induce a lack of motor reaction to stimuli and to obtain an explicit amnesia. Some studies found that general anesthesia as an independent risk factor could result in a desynchronization of the circadian time structure and cause postoperative sleep disorders characterized by reduced rapid eye movement (REM) and slow wave sleep (SWS), which have signiﬁcant deleterious impacts on postoperative outcomes, such as postoperative fatigue, severe anxiety and depression, emotional detachment and delirium, and even pain sensitivity or postoperative pain of patients.Several studies also indicated that circadian rhythms existed in human and controlled by a main internal central clock, the suprachiasmatic nuclei, located in the anterior hypothalamus, which produce and regulate biological rhythms such as sleep arousal, hormones and metabolism could also affect the dose of general anesthesics, which lead to different postoperative recoveries and may have different effects on postoperative sleep quality. Previous studies proved that postoperative sleep disturbances and poor sleep quality are associated with higher postoperative pain, changes in behavior and poor emotional well-being, which could further aggravate postoperative sleep quality. At present, there are few studies which are about the effect of circadian rhythm for different timing of surgery on intraoperative anesthestic requirement, postoperative sleep quality and pain under general anesthesia.

DETAILED DESCRIPTION:
eighty-four patients scheduled for elective laparoscopic abdominal surgeries under general anesthesia were randomly assigned to receive operation in the Day Group (8:00-12:00) and the Night Group (18:00-22:00). The Portable Sleep Monitor (PSM) was performed on the following 3 nights: the night before surgery (Sleep1), the ﬁrst night after surgery (Sleep 2), and the third night after surgery (Sleep 3). Postoperative pain scores using visual analogue scoring scale, subjective sleep quality using the Athens Insomnia Scale, total dose of general anesthetics and postoperative adverse effect were also recorded

ELIGIBILITY:
Inclusion Criteria:

* age between 18 and 65 years
* American Society of Anaesthesiologists (ASA) physical status I or II.

Exclusion Criteria:

* cardiovascular disease
* long term use of analgesic
* preoperative heart rate (HR) less than 50 beats/min
* second- or third-degree atrioventricular block
* sleep disorder
* sleep apnea syndrome
* history of abnormal operation or anesthesia recovery psychosis or a patient with a language communication disorder did not provide informed consent

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Actual)
Dates: Start 2019-09-20 (Actual); Primary Completion 2020-01-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
postoperative sleep quality of one night before surgery | one night before the surgery
  Use sleep monitor to test the sleep quality one night before surgery
postoperative sleep quality of the first night after surgery | the first night after surgery
  Use sleep monitor to test the sleep quality the first night after surgery
postoperative sleep quality of the third night after surgery | the third night after surgery
  Use sleep monitor to test the sleep quality the third night after surgery

SECONDARY OUTCOMES:
intraoperative general anesthestic requirement | during the surgery
  record the total dose of general anesthestic requirement during the operation
postoperative adverse effect | 24 hours after the surgery
  record the postoperative adverse effect

CONTACTS AND LOCATIONS:
Overall Officials: Junchao Zhu, Study Director — Shengjing Hospital
Locations (1):
- Shengjing hospital of China Medical University, Shenyang, Liaoning, China